CLINICAL TRIAL: NCT04933981
Title: Mobile PCR-based Surveillance for SARS-CoV-2 to Reduce Visiting Restrictions in Nursing Homes During the COVID-19 Pandemic
Brief Title: Benefit of Expanded Surveillance of Nursing Homes During the COVID-19 Pandemic
Status: Completed | Type: Observational
Sponsor: University of Cologne (Other)
Collaborators: City Council of Cologne, Department of Public Health, NRW, Germany (Unknown); City Council of Cologne, Department of Social Affairs, Health and Environment, NRW, Germany (Unknown)
Responsible Party: Principal Investigator, Oliver Cornely, MD, Professor, Doctor, University of Cologne
Other Study IDs: 3S fuer Koeln
Record Dates: First submitted 2021-05-21; First posted 2021-06-22 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: COVID-19 Respiratory Infection; SARS-CoV-2 Infection
Keywords: Surveillance; COVID-19 pandemic; nursing homes; visiting restrictions during the COVID-19 pandemic
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Testing for SARS-CoV-2 is performed by nasal and/or pharyngeal swab using conventional swab materials. The oropharynx and/or nasopharynx of the participants will be swabbed in an arc for approx. 5 seconds to ensure the highest possible quality of the swab.
  The swabbing is performed by qualified medical personnel using personal protective equipment including gloves, disposable gown, hood, goggles and FFP masks.
  Samples are brought to the testing laboratory within 12 hours of collection. Further analysis of the nose/throat swabs is performed by PCR at the Institute of Virology, University of Cologne.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- interventional nursing home (INH).: regular, twice to three times weekly, and voluntary, i.e. non-mandatory, on-site testing for SARS-CoV-2 of HCW and visitors (INH)
  Interventions: Diagnostic Test: Nasopharyngeal swab for SARS-CoV-2
- control nursing home (CNH): routine setting without frequent regular testing for SARS-CoV-2 (control nursing homes; CNH). Testing only performed by local health authorities upon medical indication, i.e. non-surveillance testing

INTERVENTIONS:
Diagnostic Test: Nasopharyngeal swab for SARS-CoV-2 — in the interventional group, regular, i.e. twice to three times weekly, SARS-CoV-2 testing was offered to health-care workers and visitors of nursing homes
  Groups: interventional nursing home (INH).

SUMMARY:
Residents in nursing homes for the senior citizens (NH) are at high risk for death from COVID-19. We investigated whether repeated non-mandatory RT-PCR SARS-CoV-2 surveillance of NH staff and visitors reduces COVID-19 incidence rates in NH residents and allows to reduce visiting restrictions.

DETAILED DESCRIPTION:
Nursing homes for senior citizens are considered risk areas for the transmission of SARS-CoV-2. To protect these risk groups, different strategies have been implemented within the framework of legally applicable conditions. The aim of this study is to observe two procedural standards (e.g. visiting restrictions, hygiene measurements):

* On the one hand, a standard procedure without testing of visitors and employees and
* on the other hand, a standard procedure with additional surveillance by voluntary testing of visitors and staff for SARS-CoV-2 and associated relaxation of measures for contact of visitors with residents.

Both standard procedures are designed to ensure adequate protection against infection. The standard procedure with the use of relaxing the measures after testing aims to make the experience of social isolation more bearable for the residents of care facilities and thus less stressful from a psychological point of view. The extent of such possible effects is not the subject of the present study.

The primary aim of the study is to observe the number of SARS-CoV-2 infections among residents of nursing homes for senior citizens under different procedural standards for infection control.

In this study, various measures specified by care institutions for visits to senior citizens' homes are accompanied by scientific screening. The aim of the screening and the analysis of infection protection measures is to enable this vulnerable group to regain participation in society but still slow down the spread of the virus and prevent an outbreak.

The (mobile) infection control center ("Coronamobil") of the University Hospital of Cologne (UKK) makes a decisive contribution to the longitudinal investigation of a risk population and to the early detection of chains of infection in addition to the surveillance carried out by the authorities. In this study, the Coronamobil and personnel are provided to avoid an additional screening burden for the homes.

Surveillance of nursing homes allows protection of particularly vulnerable populations in the SARS-CoV-2 pandemic, and additional controlled contact. An evidence-based, safe and human visit concept could be transferred from Cologne to the whole of Germany. The resulting scientific knowledge would additionally provide a foundation for the control of future outbreak situations.

ELIGIBILITY:
Inclusion Criteria:

* One-time or frequent visitors in care facilities of the INH group who want to be tested for SARS-CoV-2 voluntarily
* employees (HCW) in care facilities of the INH group who want to be tested voluntarily
* Successful declaration of consent via the UKK Corona web tool

Exclusion Criteria:

* Visitors and employees in care facilities of the INH group with signs of SARS-CoV-2 infection
* No participants in the context of the study are in principle:
* one-time and frequent visitors in care facilities of the CNH group
* employees in care facilities of the CNH group
* Residents in care facilities of the CNH and the INH group

Ages: 0 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: * One-time or frequent visitors in care facilities with standard 2 who want to be tested voluntarily
  * employees in care facilities with standard 2 who want to be tested voluntarily
  * Successful declaration of consent via the UHC Corona Web Tool
Sampling Method: Probability Sample
Enrollment: 1587 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
SARS-CoV-2 infection among residents | Oct 15th until Dec 18th, 2020
  SARS-CoV-2 infection among residents in INH and CNH (proof of SARS-CoV-2 DNA on nasopharyngeal swab with or without symptoms of SARS-CoV-2 infection)

SECONDARY OUTCOMES:
SARS-CoV-2 infection among visitors and health-care workers (HCW) of INH | Oct 15th until Dec 18th, 2020
  proof of SARS-CoV-2 DNA (asymptomatic and symptomatic) on nasopharyngeal swab among visitors and HCW in INH
Comparison of sensitivity of SARS-CoV-2 rtPCR and SARS-CoV-2 rapid antigen tests | Oct 15th until Dec 18th, 2020
  Ct values in RT-PCR samples of SARS-CoV-2 PCR
Overall mortality, COVID-19 related mortality, and excess mortality | up to two weeks after study completion
  Overall mortality, COVID-19 related mortality defined as death while infected with SARS-CoV-2, and excess mortality were assessed by comparing NH mortality data of the same period in the previous year.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver A Cornely, MD, Principal Investigator — University of Cologne
Locations (1):
- University Hospital Cologne, Cologne, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No
IPD can be made available upon request

REFERENCES:
- [Derived] Stemler J, Kramer T, Dimitriou V, Wieland U, Schumacher S, Sprute R, Oberste M, Wiesmuller G, Rau H, Pieper S, Bethe U, Lehmann C, Hellmich M, Klein F, Langebartels G, Cornely OA. Mobile PCR-based surveillance for SARS-CoV-2 to reduce visiting restrictions in nursing homes during the COVID-19 pandemic: a pilot study. Infection. 2022 Jun;50(3):607-616. doi: 10.1007/s15010-021-01716-4. Epub 2021 Oct 20. PMID 34669164